CLINICAL TRIAL: NCT07338617
Title: Point of Care Ultrasound (POCUS) for Diagnosis and Treatment of Fractures in the Costal Cartilage
Status: Not yet recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Erik Öberg Westin, Principal investigator, Sahlgrenska University Hospital
Other Study IDs: 286117
Record Dates: First submitted 2025-12-15; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Rib Fracture; Cartilage Damage
Keywords: Rib Fractures; Fractures, Cartilage; Ultrasonography; Traumatology
MeSH Terms: conditions — Rib Fractures; Fractures, Cartilage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group

SUMMARY:
The goal of this observational study is to learn if combining ultrasound and CT scans can better diagnose cartilage fractures in the ribs, and to understand how finding these injuries affects treatment decisions for patients with injuries to the Chest wall.

The main questions it aims to answer are:

* Does using both ultrasound and CT scans find more costal cartilage fractures than CT scans alone?
* Does discovering costal cartilage fractures change how patients are treated, such as whether more patients receive surgery or if different fractures are repaired?
* How do costal cartilage fractures heal, and do they affect lung function, pain, or the risk of complications after surgery?

Patients with cartilage injuries will be followed up at 1, 3, and 12 months after their injury. They will be checked for pain, instability, and healing using ultrasound and sometimes CT scans. The study will also assess lung function, quality of life, and pain levels.

DETAILED DESCRIPTION:
Rib fractures occur in one tenth of patients with traumatic injuries. Our knowledge about the treatment of patients with rib fractures has increased in recent years, as interest in surgical treatment of these fractures has grown. We now know more about the healing process for both surgically and conservatively treated rib fractures than we did before. Fractures in the rib cartilage are less studied. We still know very little about how fractures in the rib cartilage heal and how to approach these fractures during surgical treatment. They are also more difficult to diagnose radiologically than fractures in the bone itself.

Computed tomography (CT) is the best radiological method for diagnosing rib fractures. CT with 3D reconstructions is also a valuable preoperative mapping tool for patients who are to undergo stabilizing surgery for rib fractures. However, CT is not as sensitive for fractures in the rib cartilage, which can therefore be missed. Ultrasound has proven to be more sensitive than CT in identifying fractures in the rib cartilage.

It is unknown whether point of care ultrasound (POCUS) performed by surgeons can identify more cartilage fractures or if this affects the treatment strategy.

The purpose of this study is to investigate whether we can find more rib fractures using POCUS in combination with CT than with CT alone. We also want to study the natural course of rib cartilage fractures using POCUS, CT, and clinical examination. We will also examine whether POCUS changes our plan for treating the patients.

The project is designed as a prospective, comparative study to evaluate a standardized protocol for POCUS for identifying cartilage injuries and for assessing radiological healing of cartilage injuries.

Adult patients treated at the Department of Surgery, Sahlgrenska University Hospital with at least one rib fracture and/or sternum fracture will be asked to participate in the study until the predetermined number of 100 patients is reached.

CT scans of included patients will be reviewed by a radiologist for the presence and extent of fractures of the sternum, cartilage, and ribs, as well as the presence of pneumothorax and/or hemothorax, lung contusion, and lung laceration.

The surgeon reviews the patient's medical record to determine if the patient meets the inclusion criteria. The surgeon then performs POCUS and documents any cartilage injuries. Afterward, the surgeon assesses the CT scan. If the surgeon notes fractures during CT review or POCUS that were not described in the radiologist's report, the CT scan is re-reviewed by the radiologist. If the fractures cannot be found during the re-review, they are considered missed. The surgeon decides during CT review whether there is an indication for surgery according to current guidelines and documents which fractures are planned to be fixed. If cartilage injuries are detected by POCUS, an assessment is made to determine whether the cartilage fractures affect the indication for surgery and/or which fractures are planned to be fixed. During surgery, the injuries that are fixed are documented.

Injuries are graded according to the Abbreviated Injury Scale (AIS), the presence of flail segment, Injury Severity Score (ISS), and New Injury Severity Score (NISS).

Demographic data on included patients are collected: age, sex, height, weight, BMI, smoking status, comorbidities (COPD, asthma, pulmonary emphysema, diabetes mellitus).

Patients with cartilage injuries are followed up at 1, 3, and 12 months after the trauma. The following data are collected at follow-up visits: clinical and radiological healing. Clinical healing means absence of tenderness or palpable and/or perceived instability over the fracture. CT and POCUS are performed after 3 months. If complete radiological healing of the chest wall is lacking, repeat CT and POCUS are performed after 12 months. Radiological healing means signs of healing on CT, divided into groups of complete healing, partial healing, and no healing according to the radiologist's assessment, as well as healing or no healing according to the surgeon's assessment during POCUS.

Other variables collected at follow-up visits are lung function measured by spirometry, quality of life estimated with EQ5D, pain estimated by opioid equivalent consumption, visual analogue scale (VAS), and a graphical representation.

The natural course of fractures in the rib cartilage is incompletely explored. Cartilage fractures can contribute to instability in the chest and are currently usually operated on with the same methods as fractures in the bone itself. Knowledge about healing time and the proportion of cartilage fractures that heal may affect the choice of treatment method and improve the patient's chance of recovery from the injuries.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients (≥18 years) treated at the Department of Surgery, Sahlgrenska University Hospital, where CT has shown at least one recent injury to the chest wall.

Exclusion Criteria:

* Patients with injuries resulting from CPR, severe head injury, spinal injury, and neurological or musculoskeletal disease affecting chest mobility will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the Department of Surgery, Sahlgrenska University Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of POCUS for injuries in rib cartilage compared to CT. | Index examination at patient inclusion.

SECONDARY OUTCOMES:
Number of participants where treatment strategy is changed upon identification of cartilage fractures not seen on CT. | Assessment made at patient inclusion.
  When cartilage injuries are detected by POCUS, an assessment is made by the surgeon to determine whether the cartilage fractures affect the indication for surgery and/or which fractures are planned to be fixed. This is a binary outcome which will be answered with "yes" or "no".
Clinical healing of fractures in the rib cartilage | 1, 3 and 12 months after patient inclusion.
  Assessment of clinical healing will be made at the follow-up visits at 1, 3 and 12 months. Fractures will be regarded as clinically healed if the patient is not sore at the fracture site and there is no palpable instability. The findings will be related to whether the patient has undergone surgical fixation of rib fractures or not.
Healing of cartilage fractures assessed with POCUS | 1, 3 and 12 months after inclusion
  At 1, 3 and 12 months follow-up healing will be assessed with POCUS. The fractures will be considered healed if there is no visible fracture line and/or movement at the fracture site. The findings will be related to whether the patient has undergone surgical fixation of rib fractures or not.
Healing of cartilage fractures assessed with CT | 3 and 12 months after patient inclusion.
  At 3 month follow-up a CT examination will be performed to determine if the fractures are healed, an additional CT examination will be performed at 12 months if healing was not seen at 3 months. Fractures will be considered completely healed if there is no visible fracture line. Fractures with visible fracture line but signs of healing such as callus will be considered partially healed. Fractures with no signs of healing will be considered non-healed. The findings will be related to whether the patient has undergone surgical fixation of rib fractures or not.
Lung function with spirometry (predicted FVC) | 1, 3 and 12 months after patient inclusion.
  Spirometry will be performed to assess whether fractures in costal cartilage affects lung function. The outcome will be predicted FVC.
To what extent do costal cartilage fractures cause pain? (opioid consumption) | 1, 3 and 12 months after patient inclusion.
  Pain will be estimated with opioid equivalent consumption.
To what extent do costal cartilage fractures cause pain? (visual analogue scale) | 1, 3 and 12 months after patient inclusion.
  Pain will be estimated with a visual analogue scale.
To what extent do costal cartilage fractures cause pain? (graphical representation) | 1, 3 and 12 months after patient inclusion.
  Pain will be estimated with a graphical representation of the human body where areas of pain can be marked by the participant.
What are the complications of fixation of costal cartilage injuries? | 1, 3 and 12 months after patient inclusion.
  What is the incidence of complications of surgical fixation of rib fractures, for instance infection and osteosynthesis failure.

CONTACTS AND LOCATIONS:
Overall Officials: Eva-Corina Caragounis, Ph. D., Ass. Prof., Study Director — Institution of Clinical Sciences, Sahlgrenska Academy, Gothenburg University. Department of Surgery, Sahlgrenska University Hospital.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ziegler DW, Agarwal NN. The morbidity and mortality of rib fractures. J Trauma. 1994 Dec;37(6):975-9. doi: 10.1097/00005373-199412000-00018. PMID 7996614
- [Background] Sirmali M, Turut H, Topcu S, Gulhan E, Yazici U, Kaya S, Tastepe I. A comprehensive analysis of traumatic rib fractures: morbidity, mortality and management. Eur J Cardiothorac Surg. 2003 Jul;24(1):133-8. doi: 10.1016/s1010-7940(03)00256-2. PMID 12853057
- [Background] Ciraulo DL, Elliott D, Mitchell KA, Rodriguez A. Flail chest as a marker for significant injuries. J Am Coll Surg. 1994 May;178(5):466-70. PMID 8167883
- [Background] Tanaka H, Yukioka T, Yamaguti Y, Shimizu S, Goto H, Matsuda H, Shimazaki S. Surgical stabilization of internal pneumatic stabilization? A prospective randomized study of management of severe flail chest patients. J Trauma. 2002 Apr;52(4):727-32; discussion 732. doi: 10.1097/00005373-200204000-00020. PMID 11956391
- [Background] Granetzny A, Abd El-Aal M, Emam E, Shalaby A, Boseila A. Surgical versus conservative treatment of flail chest. Evaluation of the pulmonary status. Interact Cardiovasc Thorac Surg. 2005 Dec;4(6):583-7. doi: 10.1510/icvts.2005.111807. Epub 2005 Sep 15. PMID 17670487
- [Background] Marasco SF, Davies AR, Cooper J, Varma D, Bennett V, Nevill R, Lee G, Bailey M, Fitzgerald M. Prospective randomized controlled trial of operative rib fixation in traumatic flail chest. J Am Coll Surg. 2013 May;216(5):924-32. doi: 10.1016/j.jamcollsurg.2012.12.024. Epub 2013 Feb 13. PMID 23415550
- [Background] Liu T, Liu P, Chen J, Xie J, Yang F, Liao Y. A Randomized Controlled Trial of Surgical Rib Fixation in Polytrauma Patients With Flail Chest. J Surg Res. 2019 Oct;242:223-230. doi: 10.1016/j.jss.2019.04.005. Epub 2019 May 14. PMID 31100568
- [Background] Bottlang M, Long WB, Phelan D, Fielder D, Madey SM. Surgical stabilization of flail chest injuries with MatrixRIB implants: a prospective observational study. Injury. 2013 Feb;44(2):232-8. doi: 10.1016/j.injury.2012.08.011. Epub 2012 Aug 19. PMID 22910817
- [Background] Granhed HP, Pazooki D. A feasibility study of 60 consecutive patients operated for unstable thoracic cage. J Trauma Manag Outcomes. 2014 Dec 30;8(1):20. doi: 10.1186/s13032-014-0020-z. eCollection 2014. PMID 25642282
- [Background] Gasparri MG, Tisol WB, Haasler GB. Rib stabilization: lessons learned. Eur J Trauma Emerg Surg. 2010 Oct;36(5):435-40. doi: 10.1007/s00068-010-0048-3. Epub 2010 Sep 24. PMID 26816224
- [Background] Marasco S, Saxena P. Surgical rib fixation - technical aspects. Injury. 2015 May;46(5):929-32. doi: 10.1016/j.injury.2014.12.021. Epub 2015 Jan 10. PMID 25624272
- [Background] Schulz-Drost S, Grupp S, Pachowsky M, Oppel P, Krinner S, Mauerer A, Hennig FF, Langenbach A. Stabilization of flail chest injuries: minimized approach techniques to treat the core of instability. Eur J Trauma Emerg Surg. 2017 Apr;43(2):169-178. doi: 10.1007/s00068-016-0664-7. Epub 2016 Mar 22. PMID 27084543
- [Background] Bauman ZM, Beard R, Cemaj S. When less is more: A minimally invasive, intrathoracic approach to surgical stabilization of rib fractures. Trauma Case Rep. 2021 Mar 11;32:100452. doi: 10.1016/j.tcr.2021.100452. eCollection 2021 Apr. PMID 33778146
- [Background] Pieracci FM, Johnson JL, Stovall RT, Jurkovich GJ. Completely thoracoscopic, intra-pleural reduction and fixation of severe rib fractures. Trauma Case Rep. 2015 Nov 4;1(5-8):39-43. doi: 10.1016/j.tcr.2015.10.001. eCollection 2015 Oct. No abstract available. PMID 30101174
- [Background] Zhang J, Hong Q, Mo X, Ma C. Complete Video-assisted Thoracoscopic Surgery for Rib Fractures: Series of 35 Cases. Ann Thorac Surg. 2022 Feb;113(2):452-458. doi: 10.1016/j.athoracsur.2021.01.065. Epub 2021 Mar 3. PMID 33675706
- [Background] Nowack T, Nonnemacher C, Christie DB. Video-Assisted Thoracoscopic Surgery as an Adjunct to Rib Fixation. Am Surg. 2022 Jun;88(6):1338-1340. doi: 10.1177/0003134820943642. Epub 2020 Aug 26. No abstract available. PMID 32845731
- [Background] Fraser SF, Tan C, Kuppusamy MK, Gukop P, Hunt IJ. The role of a video-assisted thoracic approach for rib fixation. Eur J Trauma Emerg Surg. 2017 Apr;43(2):185-190. doi: 10.1007/s00068-016-0641-1. Epub 2016 Feb 5. PMID 26850079
- [Background] Xia H, Zhu P, Li J, Zhu D, Sun Z, Deng L, Zhang Y, Wang D. Thoracoscope combined with internal support system of chest wall in open reduction and internal fixation for multiple rib fractures. Exp Ther Med. 2018 Dec;16(6):4650-4654. doi: 10.3892/etm.2018.6817. Epub 2018 Oct 1. PMID 30542416
- [Background] Oberg Westin E, Fagevik Olsen M, Ortenwall P, Caragounis EC. Retrospective comparison of operative technique for chest wall injuries. Injury. 2023 Mar 10:S0020-1383(23)00248-6. doi: 10.1016/j.injury.2023.03.012. Online ahead of print. PMID 36925375
- [Background] Tay-Lasso E, Alaniz L, Grant W, Hovis G, Frank M, Kincaid C, Brynn S, Pieracci FM, Nahmias J, Barrios C, Rockne W, Chin T, Swentek L, Schubl SD. Prospective single-center paradigm shift of surgical stabilization of rib fractures with decreased length of stay and operative time with an intrathoracic approach. J Trauma Acute Care Surg. 2023 Apr 1;94(4):567-572. doi: 10.1097/TA.0000000000003811. Epub 2022 Oct 25. PMID 36301075
- [Background] Tichenor M, Reparaz LB, Watson C, Reeves J, Prest P, Fitzgerald M, Patel N, Tan X, Hessey J. Intrathoracic plates versus extrathoracic plates: a comparison of postoperative pain in surgical stabilization of rib fracture technique. Trauma Surg Acute Care Open. 2023 Nov 3;8(1):e001201. doi: 10.1136/tsaco-2023-001201. eCollection 2023. PMID 37936903
- [Background] Marasco S, Liew S, Edwards E, Varma D, Summerhayes R. Analysis of bone healing in flail chest injury: do we need to fix both fractures per rib? J Trauma Acute Care Surg. 2014 Sep;77(3):452-8. doi: 10.1097/TA.0000000000000375. PMID 25159250
- [Background] Pishbin E, Ahmadi K, Foogardi M, Salehi M, Seilanian Toosi F, Rahimi-Movaghar V. Comparison of ultrasonography and radiography in diagnosis of rib fractures. Chin J Traumatol. 2017 Aug;20(4):226-228. doi: 10.1016/j.cjtee.2016.04.010. Epub 2017 May 26. PMID 28687342
- [Background] Sano A. Rib Radiography versus Chest Computed Tomography in the Diagnosis of Rib Fractures. Thorac Cardiovasc Surg. 2018 Nov;66(8):693-696. doi: 10.1055/s-0038-1645887. Epub 2018 May 1. PMID 29715707
- [Background] Lee WS, Kim YH, Chee HK, Lee SA. Ultrasonographic evaluation of costal cartilage fractures unnoticed by the conventional radiographic study and multidetector computed tomography. Eur J Trauma Emerg Surg. 2012 Feb;38(1):37-42. doi: 10.1007/s00068-011-0117-2. Epub 2011 May 25. PMID 26815671
- [Background] Nummela MT, Bensch FV, Pyhalto TT, Koskinen SK. Incidence and Imaging Findings of Costal Cartilage Fractures in Patients with Blunt Chest Trauma: A Retrospective Review of 1461 Consecutive Whole-Body CT Examinations for Trauma. Radiology. 2018 Feb;286(2):696-704. doi: 10.1148/radiol.2017162429. Epub 2017 Nov 2. PMID 29095676
- [Background] Sermonesi G, Bertelli R, Pieracci FM, Balogh ZJ, Coimbra R, Galante JM, Hecker A, Weber D, Bauman ZM, Kartiko S, Patel B, Whitbeck SS, White TW, Harrell KN, Perrina D, Rampini A, Tian B, Amico F, Beka SG, Bonavina L, Ceresoli M, Cobianchi L, Coccolini F, Cui Y, Dal Mas F, De Simone B, Di Carlo I, Di Saverio S, Dogjani A, Fette A, Fraga GP, Gomes CA, Khan JS, Kirkpatrick AW, Kruger VF, Leppaniemi A, Litvin A, Mingoli A, Navarro DC, Passera E, Pisano M, Podda M, Russo E, Sakakushev B, Santonastaso D, Sartelli M, Shelat VG, Tan E, Wani I, Abu-Zidan FM, Biffl WL, Civil I, Latifi R, Marzi I, Picetti E, Pikoulis M, Agnoletti V, Bravi F, Vallicelli C, Ansaloni L, Moore EE, Catena F. Surgical stabilization of rib fractures (SSRF): the WSES and CWIS position paper. World J Emerg Surg. 2024 Oct 18;19(1):33. doi: 10.1186/s13017-024-00559-2. PMID 39425134